CLINICAL TRIAL: NCT01945398
Title: Effect of Inspiratory Muscle Training in the Ventilatory Muscle Metaboreflex in Chronic Obstructive Pulmonary Disease Patients.
Brief Title: IMT in Ventilatory Muscle Metaboreflex in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Danilo C Berton, MD, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 120489
Record Dates: First submitted 2013-09-15; First posted 2013-09-18 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Pulmonary Rehabilitation; Inspiratory Muscle Training; Inspiratory Muscle Strength; Vascular Resistance; Exercise; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inspiratory Muscle Training (IMT) (Experimental): Patients from the inspiratory muscle training group will utilize a linear pressoric resistance equipment with an inspiratory charge of 30% of maximum inspiratory pressure (adjusted weekly), during 7 days of the week, session duration of 30 minutes, during 8 weeks.
  Interventions: Other: Inspiratory Muscle Training
- Sham IMT (Placebo Comparator): Patients in the placebo group will be submitted to inspiratory muscle training with the same equipment as the intervention group, however without a resistance generating spring.
  Interventions: Other: SHAM

INTERVENTIONS:
Other: Inspiratory Muscle Training — Patients will receive IMT for 30 min, 7 times per week, for 8 weeks using Inspiratory Muscle Trainer device (PowerBreath Inc.). During training, patients will be instructed to maintain diaphragmatic breathing, with a breathing rate at 15 to 20 breaths/min. Inspiratory load was set at 30% of maximal static inspiratory pressure, and weekly training loads were adjusted to maintain 30% of the PImax. Each week, six training sessions were performed at home and one training session was supervised at the hospital.
  Arms: Inspiratory Muscle Training (IMT)
Other: SHAM — Patients will receive SHAM training for 30 min, 7 times per week, for 8 weeks using Inspiratory Muscle Trainer device (PowerBreath Inc.) without load. Patients will be instructed to maintain diaphragmatic breathing, with a breathing rate at 15 to 20 breaths/min. Each week, six training sessions were performed at home and one training session was supervised at the hospital.
  Arms: Sham IMT

SUMMARY:
This research intends to evaluate if inspiratory muscle training (IMT) reduces inspiratory muscle metaboreflex through the decrease of calf vascular resistance and increase of calf blood flow in Chronic Obstructive Pulmonary Disease (COPD).

DETAILED DESCRIPTION:
Patients will be selected from the Hospital de Clinicas de Porto Alegre's COPD ambulatory, by convenience. Afterwards, patients will be submitted to pulmonary function test (spirometry) and cardiopulmonary exercise tests (incremental and submaximal), maximal inspiratory pressure evaluation and induction of the inspiratory muscle metaboreflex through venous occlusion plethysmography. Disease specific health related quality of life questionnaire (Saint George Respiratory Questionnaire) and daily life dyspnea questionnaire (Baseline Dyspnea Index and Transitional Dyspnea Index) will be administered at the first and last visit of each subject. Patients will undergo inspiratory muscle training for 30 minutes per day, 7 times a week, for 8 weeks, with Inspiratory Muscle Trainer device (PowerBreath Inc.). There will be a weekly follow up at the institution's Clinical Research Center, where maximal inspiratory pressure (PImax) and inspiratory training techniques will be reevaluated. After this period, tests of pulmonary function, questionnaires exercise tolerance and induction of the inspiratory muscle metaboreflex will be reevaluated.

ELIGIBILITY:
Inclusion Criteria:

Selection of subjects will be made through the Hospital de Clinicas de Porto Alegre Pneumology Service's COPD ambulatory. The inclusion criteria consist of -patients with COPD with functional confirmation through spirometry as by previously defined criteria.

Those selected must be classified as GOLD II-IV, with moderate to severe expiratory flow obstruction.

Exclusion Criteria:

Patients will be considered ineligible for this study if they

* develop COPD exacerbation 8 weeks prior to recruitment
* if systemic corticosteroids are utilized (in the last three months)
* if there is history of acute myocardial infarction (in the last three months)
* if there is presence of neuromuscular disease
* history of cardiovascular disease or active smoking (in the last 6 months)
* clinical history of peripheral vascular disease and if age is equal or superior to 85 years

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Calf blood flow | 8 weeks

SECONDARY OUTCOMES:
Time to exercise tolerance (tlim) | 8 weeks
  Exercise time during high intensity submaximal Cardiopulmonary exercise testing
Maximum Inspiratory Pressure | 8 weeks
The St George's Respiratory Questionnaire | 8 weeks
Baseline Dyspnea Index/Transitional Dyspnea Index | 8 weeks
Calf vascular resistance | 8 weeks
  Calf blood flow/mean arterial pressure

CONTACTS AND LOCATIONS:
Overall Officials: Danilo C Berton, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Background] Rabe KF, Hurd S, Anzueto A, Barnes PJ, Buist SA, Calverley P, Fukuchi Y, Jenkins C, Rodriguez-Roisin R, van Weel C, Zielinski J; Global Initiative for Chronic Obstructive Lung Disease. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2007 Sep 15;176(6):532-55. doi: 10.1164/rccm.200703-456SO. Epub 2007 May 16. PMID 17507545
- [Background] Aliverti A, Macklem PT. The major limitation to exercise performance in COPD is inadequate energy supply to the respiratory and locomotor muscles. J Appl Physiol (1985). 2008 Aug;105(2):749-51; discussion 755-7. doi: 10.1152/japplphysiol.90336.2008. Epub 2008 Mar 20. No abstract available. PMID 18678622
- [Background] Debigare R, Maltais F. The major limitation to exercise performance in COPD is lower limb muscle dysfunction. J Appl Physiol (1985). 2008 Aug;105(2):751-3; discussion 755-7. doi: 10.1152/japplphysiol.90336.2008a. No abstract available. PMID 18678623
- [Background] O'Donnell DE, Webb KA. The major limitation to exercise performance in COPD is dynamic hyperinflation. J Appl Physiol (1985). 2008 Aug;105(2):753-5; discussion 755-7. doi: 10.1152/japplphysiol.90336.2008b. No abstract available. PMID 18678624
- [Background] Neder JA, Jones PW, Nery LE, Whipp BJ. Determinants of the exercise endurance capacity in patients with chronic obstructive pulmonary disease. The power-duration relationship. Am J Respir Crit Care Med. 2000 Aug;162(2 Pt 1):497-504. doi: 10.1164/ajrccm.162.2.9907122. PMID 10934077
- [Background] Puente-Maestu L, Garcia de Pedro J, Martinez-Abad Y, Ruiz de Ona JM, Llorente D, Cubillo JM. Dyspnea, ventilatory pattern, and changes in dynamic hyperinflation related to the intensity of constant work rate exercise in COPD. Chest. 2005 Aug;128(2):651-6. doi: 10.1378/chest.128.2.651. PMID 16100150
- [Background] Chiappa GR, Borghi-Silva A, Ferreira LF, Carrascosa C, Oliveira CC, Maia J, Gimenes AC, Queiroga F Jr, Berton D, Ferreira EM, Nery LE, Neder JA. Kinetics of muscle deoxygenation are accelerated at the onset of heavy-intensity exercise in patients with COPD: relationship to central cardiovascular dynamics. J Appl Physiol (1985). 2008 May;104(5):1341-50. doi: 10.1152/japplphysiol.01364.2007. Epub 2008 Mar 20. PMID 18356477
- [Background] Neder JA. The major limitation to exercise performance in COPD is inadequate energy supply to the respiratory and locomotor muscles vs. lower limb muscle dysfunction vs. dynamic hyperinflation. Interpretation of exercise intolerance in COPD requires an integrated, multisystemic approach. J Appl Physiol (1985). 2008 Aug;105(2):758-9. doi: 10.1152/japplphysiol.90336.2008e. No abstract available. PMID 18678626
- [Background] Nici L, Donner C, Wouters E, Zuwallack R, Ambrosino N, Bourbeau J, Carone M, Celli B, Engelen M, Fahy B, Garvey C, Goldstein R, Gosselink R, Lareau S, MacIntyre N, Maltais F, Morgan M, O'Donnell D, Prefault C, Reardon J, Rochester C, Schols A, Singh S, Troosters T; ATS/ERS Pulmonary Rehabilitation Writing Committee. American Thoracic Society/European Respiratory Society statement on pulmonary rehabilitation. Am J Respir Crit Care Med. 2006 Jun 15;173(12):1390-413. doi: 10.1164/rccm.200508-1211ST. No abstract available. PMID 16760357
- [Background] Gayan-Ramirez G, Koulouris N, Roca J, Decramer M. Respiratory and skeletal muscles in chronic obstructive pulmonary disease. Eur Respir Mon 2006; 38: 201-223.
- [Background] St Croix CM, Morgan BJ, Wetter TJ, Dempsey JA. Fatiguing inspiratory muscle work causes reflex sympathetic activation in humans. J Physiol. 2000 Dec 1;529 Pt 2(Pt 2):493-504. doi: 10.1111/j.1469-7793.2000.00493.x. PMID 11101657
- [Background] Harms CA, Babcock MA, McClaran SR, Pegelow DF, Nickele GA, Nelson WB, Dempsey JA. Respiratory muscle work compromises leg blood flow during maximal exercise. J Appl Physiol (1985). 1997 May;82(5):1573-83. doi: 10.1152/jappl.1997.82.5.1573. PMID 9134907
- [Background] Sheel AW, Derchak PA, Morgan BJ, Pegelow DF, Jacques AJ, Dempsey JA. Fatiguing inspiratory muscle work causes reflex reduction in resting leg blood flow in humans. J Physiol. 2001 Nov 15;537(Pt 1):277-89. doi: 10.1111/j.1469-7793.2001.0277k.x. PMID 11711580
- [Background] Dempsey JA, Romer L, Rodman J, Miller J, Smith C. Consequences of exercise-induced respiratory muscle work. Respir Physiol Neurobiol. 2006 Apr 28;151(2-3):242-50. doi: 10.1016/j.resp.2005.12.015. PMID 16616716
- [Background] Levison H, Cherniack RM. Ventilatory cost of exercise in chronic obstructive pulmonary disease. J Appl Physiol. 1968 Jul;25(1):21-7. doi: 10.1152/jappl.1968.25.1.21. No abstract available. PMID 5661150
- [Background] Aliverti A, Macklem PT. How and why exercise is impaired in COPD. Respiration. 2001;68(3):229-39. doi: 10.1159/000050502. PMID 11416240
- [Background] Borghi-Silva A, Oliveira CC, Carrascosa C, Maia J, Berton DC, Queiroga F Jr, Ferreira EM, Almeida DR, Nery LE, Neder JA. Respiratory muscle unloading improves leg muscle oxygenation during exercise in patients with COPD. Thorax. 2008 Oct;63(10):910-5. doi: 10.1136/thx.2007.090167. Epub 2008 May 20. PMID 18492743
- [Background] Chiappa GR, Queiroga F Jr, Meda E, Ferreira LF, Diefenthaeler F, Nunes M, Vaz MA, Machado MC, Nery LE, Neder JA. Heliox improves oxygen delivery and utilization during dynamic exercise in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2009 Jun 1;179(11):1004-10. doi: 10.1164/rccm.200811-1793OC. Epub 2009 Mar 19. PMID 19299497
- [Background] Berton DC, Barbosa PB, Takara LS, Chiappa GR, Siqueira AC, Bravo DM, Ferreira LF, Neder JA. Bronchodilators accelerate the dynamics of muscle O2 delivery and utilisation during exercise in COPD. Thorax. 2010 Jul;65(7):588-93. doi: 10.1136/thx.2009.120857. PMID 20627914
- [Background] Mancini D, Donchez L, Levine S. Acute unloading of the work of breathing extends exercise duration in patients with heart failure. J Am Coll Cardiol. 1997 Mar 1;29(3):590-6. doi: 10.1016/s0735-1097(96)00556-6. PMID 9060898
- [Background] O'Donnell DE, D'Arsigny C, Raj S, Abdollah H, Webb KA. Ventilatory assistance improves exercise endurance in stable congestive heart failure. Am J Respir Crit Care Med. 1999 Dec;160(6):1804-11. doi: 10.1164/ajrccm.160.6.9808134. PMID 10588589
- [Background] Chiappa GR, Roseguini BT, Vieira PJ, Alves CN, Tavares A, Winkelmann ER, Ferlin EL, Stein R, Ribeiro JP. Inspiratory muscle training improves blood flow to resting and exercising limbs in patients with chronic heart failure. J Am Coll Cardiol. 2008 Apr 29;51(17):1663-71. doi: 10.1016/j.jacc.2007.12.045. PMID 18436118
- [Background] McConnell AK, Lomax M. The influence of inspiratory muscle work history and specific inspiratory muscle training upon human limb muscle fatigue. J Physiol. 2006 Nov 15;577(Pt 1):445-57. doi: 10.1113/jphysiol.2006.117614. Epub 2006 Sep 14. PMID 16973699
- [Background] Witt JD, Guenette JA, Rupert JL, McKenzie DC, Sheel AW. Inspiratory muscle training attenuates the human respiratory muscle metaboreflex. J Physiol. 2007 Nov 1;584(Pt 3):1019-28. doi: 10.1113/jphysiol.2007.140855. Epub 2007 Sep 13. PMID 17855758
- [Background] Troosters T, Gosselink R, Decramer M. Chronic obstructive pulmonary disease and chronic heart failure: two muscle diseases? J Cardiopulm Rehabil. 2004 May-Jun;24(3):137-45. doi: 10.1097/00008483-200405000-00001. PMID 15235292
- [Background] Muthumala A. Chronic heart failure and chronic obstructive pulmonary disease: one problem, one solution? Int J Cardiol. 2008 Mar 28;125(1):1-3. doi: 10.1016/j.ijcard.2007.07.160. Epub 2007 Nov 26. PMID 18035433
- [Background] Gosselink R, De Vos J, van den Heuvel SP, Segers J, Decramer M, Kwakkel G. Impact of inspiratory muscle training in patients with COPD: what is the evidence? Eur Respir J. 2011 Feb;37(2):416-25. doi: 10.1183/09031936.00031810. PMID 21282809
- [Background] Dall'Ago P, Chiappa GR, Guths H, Stein R, Ribeiro JP. Inspiratory muscle training in patients with heart failure and inspiratory muscle weakness: a randomized trial. J Am Coll Cardiol. 2006 Feb 21;47(4):757-63. doi: 10.1016/j.jacc.2005.09.052. Epub 2006 Jan 26. PMID 16487841
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Pereira CA, Sato T, Rodrigues SC. New reference values for forced spirometry in white adults in Brazil. J Bras Pneumol. 2007 Jul-Aug;33(4):397-406. doi: 10.1590/s1806-37132007000400008. English, Portuguese. PMID 17982531
- [Background] Orsted HC, Baerentsen K, Jensen VG, Kofod H, Thorn NA, Trolle D. [On the origin and benefits of amniotic fluid. [Reprint of 1797 edition]. Published with comments and notes by the Danish society of the history of pharmacy. With historical contributions by K. Baerentsen, V. G. Jensen, H. Kofod, N. A. Thorn, D. Trolle]. Theriaca. 1977;18:1-107. No abstract available. Danish. PMID 11633911
- [Background] Neder JA, Andreoni S, Castelo-Filho A, Nery LE. Reference values for lung function tests. I. Static volumes. Braz J Med Biol Res. 1999 Jun;32(6):703-17. doi: 10.1590/s0100-879x1999000600006. PMID 10412549
- [Background] Neder JA, Andreoni S, Peres C, Nery LE. Reference values for lung function tests. III. Carbon monoxide diffusing capacity (transfer factor). Braz J Med Biol Res. 1999 Jun;32(6):729-37. doi: 10.1590/s0100-879x1999000600008. PMID 10412551
- [Background] Neder JA, Andreoni S, Lerario MC, Nery LE. Reference values for lung function tests. II. Maximal respiratory pressures and voluntary ventilation. Braz J Med Biol Res. 1999 Jun;32(6):719-27. doi: 10.1590/s0100-879x1999000600007. PMID 10412550